CLINICAL TRIAL: NCT03129698
Title: Phase II Study of Apatinib in Maintenance Treatment of Extensive-stage Small-cell Lung Cancer
Brief Title: The Efficacy and Safety of Apatinib Monotherapy in Maintenance Treatment of Extensive-stage Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junling Li (Other)
Responsible Party: Sponsor-Investigator, Junling Li, Clinical Professor, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-066-SL
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Apatinib in Maintenance Treatment
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Patients with untreated extensive-stage small-cell lung cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formerly Arm Label (Other): Apatinib 250mg daily
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 250mg daily

SUMMARY:
52 patients with extensive-stage small-cell lung cancer and without progression after completing chemotherapy, will receive apatinib monotherapy as maintenance therapy.

DETAILED DESCRIPTION:
52 patients with extensive-stage small-cell lung cancer, who had a best response of complete response (CR), partial response (PR), or stable disease (SD) after completing chemotherapy will receive apatinib monotherapy as maintenance therapy after chemotherapy to evaluate the efficacy and safety of maintenance apatinib after chemotherapy for small-cell lung cancer. At the same time, we will explore the correlation between efficacy and tumor stem cell markers expression by taking peripheral blood to detect tumor stem cell markers. The primary end point is progression-free survival (PFS). The secondary end point is overall survival (OS), toxicity, and the correlation between efficacy and tumor stem cell markers expression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small-cell lung cancer and extensive stage (extrathoracic metastatic disease, malignant pleural effusion, contralateral supraclavicular adenopathy, or contralateral hilar adenopathy)
* Having a best response of complete response (CR), partial response (PR), or stable disease (SD) after completing chemotherapy, or combining sequential radiotherapy
* Prior treatment without c-kit targeted drugs
* Life expectancy of more than 3 months
* Age ≥ 18 years
* Oncology Group performance status of 0 to 2
* Informed consent.

Exclusion Criteria:

* Mixed lung cancer or other types of lung cancer
* Have previously received c-kit targeted drugs
* Hemoglobin<8.0 g/dL, white blood cell <3 X 10^9/L, platelet count <75 X 10^9/L, alanine aminotransferase, glutamic-oxalacetic transaminase, blood urine nitrogen and creatinine more than normal limits on 3.0 times
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Patients had recent major surgery, significant hemoptysis ( 5 ml), open wounds, or brain metastases present on required pre-enrollment brain imaging or required full-dose anticoagulation
* Uncontrol hypertension, >160/100 mmHg after treatment
* Pregnant or lactating patients
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) infection
* Patients who are suffering from serious autoimmune disease
* Patients who had active infection
* Patients who are suffering from serious organ dysfunction
* Patients who are suffering from other cancer
* Other situations that the researchers considered unsuitable for this study.
* Other concurrent uncontrolled illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months

SECONDARY OUTCOMES:
Number of participants with Adverse events | 6 months
  Drug related side effects
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Junling Li, Beijing, Beijing Municipality, China